CLINICAL TRIAL: NCT01856777
Title: Evaluating the Effectiveness of Pregnancy Tests as an Assessment Tool to Identify Continuing Pregnancy After Early Medical Abortion
Brief Title: Effectiveness of Pregnancy Tests as an Assessment Tool to Identify Continuing Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 6003
Record Dates: First submitted 2013-05-03; First posted 2013-05-17 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Medical Abortion
Keywords: Medical Abortion; Pregnancy Test; continuing pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High sensitivity urine pregnancy test (Other): Standard medical care and high sensitivity urine pregnancy test
  Interventions: Device: High sensitivity urine pregnancy test
- Semi-quantitative panel test (Other): Standard medical care and semi-quantitative panel test
  Interventions: Device: Semi-quantitative panel test

INTERVENTIONS:
Device: Semi-quantitative panel test
  Other Names: dBest (AmeriTek, Seattle WA, USA)
  Arms: Semi-quantitative panel test
Device: High sensitivity urine pregnancy test
  Other Names: Quickstick one-step hCG Pregnancy Test, Phamatech, San Diego, CA, USA
  Arms: High sensitivity urine pregnancy test

SUMMARY:
This randomized study will examine the effectiveness of two types of pregnancy tests (a semi-quantitative test and a high sensitivity test) to identify continuing pregnancy at home at various time points after early medical abortion. The first test a semi-quantitative panel test marketed under the brand name dBest (AmeriTek, Seattle WA, USA). This urine-based, one-step kit has been used in two previous studies in Vietnam (12, 13). The second test is a locally available urine dipstick (Quickstick one-step hCG Pregnancy Test, Phamatech, San Diego, CA, USA).

1. The investigators hypothesize that 99% of the SQPT and 35% of the HSPT will correctly identify ongoing pregnancy at day 14.
2. The investigators hypothesize that 99% of the SQPT and 25% of the HSPT will correctly identify ongoing pregnancy at day 7.
3. The investigators hypothesize that 75% of the SQPT and 10% of the HSPT will correctly identify ongoing pregnancy at day 4.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤63days from LMP
* Eligible for mifepristone- misoprostol medical abortion according to clinic guidelines(national guidelines stipulate that women can receive medical abortion thru 63 days LMP at Hung Vuong (tertiary level) hospital; women with gestations up to 49 days LMP can receive medical abortion at Hocmon (district) hospital)
* Willing to follow instructions of the provider regarding use of the pregnancy tests
* Able to read and write to use pregnancy test at home
* Willing to be randomized to perform one of two types of urine pregnancy tests at three time points at home
* Willing to provide an address and/or telephone number for purposes of follow-up
* Agrees to return for follow-up visit at clinic to confirm abortion status
* Wishes to participate in the study
* Able to consent to study participation

Exclusion Criteria:

* Women not meeting the above inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of these two types of home pregnancy tests | 2 weeks
  Accuracy of these two types of home pregnancy tests to identify continuing pregnancy at four, seven and fourteen days after mifepristone administration.

SECONDARY OUTCOMES:
Comparison of the two types of pregnancy tests at identifying continuing pregnancy | 2 weeks
The use and acceptability of the two tests | 2 weeks
  The use and acceptability of the two tests for women as a diagnostic tool to assess pregnancy status at home following early medical abortion
Correlation between the pregnancy test results determined by the woman at home and the abortion outcome determined by provider | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Nguyen Thi Nhu Ngoc, MD, MsC, Principal Investigator — CRCRH; Paul Blumenthal, MD, Principal Investigator — Stanford University; Wendy Sheldon, MPH, MSW, PhD, Principal Investigator — Gynuity Health Projects
Locations (2):
- Vietnam (2):
  - Hocmon General District Hospital, Hochiminh City
  - Hungvuong Hospital, Hochiminh City